CLINICAL TRIAL: NCT00052416
Title: Thalidomide in Indolent Non-Hodgkin's Lymphoma: A Feasibility Study
Brief Title: Thalidomide in Treating Patients With Asymptomatic, Indolent Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: BIDMC-W-01-0384-FB; CDR0000258419 (Registry Identifier: PDQ (Physician Data Query)); NEDH-W-01-0384-FB; BIDMC-2001-P-001950; NCI-V02-1714
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2003-04

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage I grade 1 follicular lymphoma; stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; Waldenström macroglobulinemia; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase I trial to determine the effectiveness of thalidomide in treating patients who have asymptomatic, indolent non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility, in terms of toxicity and patient compliance, of thalidomide in patients with asymptomatic, indolent non-Hodgkin's lymphoma or chronic lymphocytic leukemia.
* Determine the event-free and progression-free survival of patients treated with this drug.
* Determine disease response and time to next treatment in patients treated with this drug.
* Determine the quality of life of patients treated with this drug.

OUTLINE: Patients receive oral thalidomide once daily. Treatment continues for 18 months in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, monthly during study, and at the end of the study.

PROJECTED ACCRUAL: A total of 30-36 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed indolent lymphoma or leukemia of one of the following subtypes:

  * Chronic lymphocytic leukemia
  * Follicular center lymphoma (grade I or II)
  * Lymphoplasmacytic lymphoma
  * Marginal zone lymphoma (nodal, extranodal, or splenic)
  * Small lymphocytic lymphoma
  * Waldenstrom's macroglobulinemia
* Any stage of disease allowed
* No hairy cell leukemia
* No T-cell lymphomas
* No prior treatment for lymphoma/leukemia
* Considered appropriate for expectant management

  * Must not require cytotoxic therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin greater than 10.0 g/dL
* Platelet count greater than 75,000/mm^3

Hepatic

* Bilirubin no greater than 2 times normal
* AST and ALT no greater than 2 times normal

Renal

* Creatinine no greater than 2.0 mg/dL

Cardiovascular

* No uncontrolled congestive heart failure
* No New York Heart Association class III or IV heart disease
* No unstable coronary artery disease
* No myocardial infarction in the past 6 months
* No serious or uncontrolled arrhythmias
* No history of thromboembolic disease

Pulmonary

* No asthma or chronic obstructive pulmonary disease requiring the use of home oxygen or frequent oral steroids (prednisone greater than 20 mg per day for 5 days within the past 3 months)

Other

* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Not planning to become pregnant in the next 2 years
* Fertile female patients must use 1 highly effective method and 1 additional effective method of contraception for 1 month prior to, during, and for 1 month after study participation
* Male patients must use effective barrier contraception during and for 1 month after study participation
* Willing and able to participate in the S.T.E.P.S. (System for Thalidomide Education and Prescribing Safety) program
* No contraindications to meeting the requirements of the S.T.E.P.S. program
* No other prior malignancy except curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix
* No peripheral neuropathy
* No poorly controlled diabetes defined by either of the following:

  * Glycosylated hemoglobin greater than 8.0 g/dL
  * Known end organ disease (i.e., nephropathy, retinopathy, or neuropathy)
* No other concurrent illness that would preclude study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Joyce, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont